CLINICAL TRIAL: NCT06158308
Title: Outcome of Laparoscopic Appendicectomy Versus Open Appendicectomy in Sudanese Patients: Cross-sectional Study
Brief Title: Outcome of Laparoscopic Appendicectomy Versus Open Appendicectomy in Sudanese Patients
Status: Completed | Type: Observational
Sponsor: National Center for Gastroentestinal and Liver Disease (Other)
Responsible Party: Sponsor
Other Study IDs: GastroentestinalLiver
Record Dates: First submitted 2023-11-18; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: General Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laparoscopic Appendicectomy
  Interventions: Procedure: Laproscopic Appendicectomy
- Open Appendicectomy
  Interventions: Procedure: Open Appendicectomy

INTERVENTIONS:
Procedure: Laproscopic Appendicectomy — A type of surgery done without a large incision. Instead, from 1 to 3 tiny cuts are made. A long, thin tube called a laparoscope is put into one of the incisions. It has a tiny video camera and surgical tools.
  Other Names: Regular surgical site dressing
  Groups: Laparoscopic Appendicectomy
Procedure: Open Appendicectomy — A cut or incision about 2 to 4 inches long is made in the lower right-hand side of your belly or abdomen. The appendix is taken out through the incision.
  Other Names: Regular surgical site dressing
  Groups: Open Appendicectomy

SUMMARY:
Background: Laparoscopic appendectomy as a minimal invasive procedure had low morbidity and mortality. It affords a direct diagnosis of the problem, allows determination of the appropriate treatment. Open appendectomy is global treatment of acute appendicitis can be done by many incisions, and associated with considerable complications.

Materials and Methods: This is a cross sectional descriptive hospital-based study to study the outcome of laparoscopic appendectomy versus open appendectomy at Elmak Nimer University Hospital over the study period. All patients in the study period who underwent appendectomy was included, data is collected through standard structured data collection sheet and analyzed by using SPSS v24.0.

ELIGIBILITY:
Inclusion Criteria:

* All patients in the study period who underwent appendectomy were included.

Exclusion Criteria:

* Patientspresented with complicated appendicitis
* Acute appendicitis with comorbiditites
* Pregnant ladies
* Patients of stump appendicitis .
* Patient with inadequate data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study includes all patients those underwent appendectomy during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2019-01-13 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
The rate of post-operative complications | Jan 2019 - Jan 2021
  the rate of postoperative complications, such as surgical site infections, intra-abdominal abscess formation, and other adverse events. The comparison would help assess the efficacy and safety of each surgical approach in the context of appendectomies.

CONTACTS AND LOCATIONS:
Locations (1):
- Medicine, Elmak Nemir University, Shandi, Alnahr Alabyad, Sudan

IPD SHARING:
Plan to Share IPD: Undecided